CLINICAL TRIAL: NCT06001567
Title: A Single-center, Single-arm Study of Avatrombopag for Patients With Hepatocellular Carcinoma and Thrombocytopenia Who Intend to Undergo Transarterial Chemoembolization and/or Hepatic Arterial Infusion Chemotherapy
Brief Title: Avatrombopag for HCC Patients With Thrombocytopenia Who Intend to Undergo TACE and/or HAIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-12
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Thrombocytopenia; Hepatocellular Carcinoma
Keywords: Thrombocytopenia; Hepatocellular Carcinoma; Transarterial Chemoembolization; hepatic arterial infusion chemotherapy
MeSH Terms: conditions — Thrombocytopenia; Carcinoma, Hepatocellular | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag (Experimental): Patients receive avatrombopag treatment 5-10 days.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag (platelet count [PLT] <40×10^9/L, 60mg P.O. QD; PLT of 40-75×10^9/L, 40mg P.O. QD) will be administered to the patients and last 5-10 days. When the PLT reaches ≥100×10^9/L, the treatment will be discontinued.

SUMMARY:
This study is conducted to evaluate the efficacy of avatrombopag for thrombocytopenia in patients with hepatocellular carcinoma (HCC) who intend to undergo transarterial chemoembolization (TACE) and/or hepatic arterial infusion chemotherapy (HAIC).

DETAILED DESCRIPTION:
This is a single-center, prospective study to evaluate the efficacy of avatrombopag for thrombocytopenia in HCC patients who intend to undergo TACE and/or HAIC.

30 HCC patients with thrombocytopenia will be enrolled in this study. Avatrombopag (platelet count [PLT] <40×10^9/L, 60mg P.O. QD; PLT of 40-75×10^9/L, 40mg P.O. QD) will be administered to the patients and last 5-10 days. When the PLT reaches ≥100×10^9/L, the treatment will be discontinued.

The primary end point of this study is the proportion of patients with PLT >75×10^9/L or doubling from baseline. The secondary endpoints are the proportion of patients with PLT >75×10^9/L, the proportion of patients with PLT doubling from baseline, the increace in PLT, the proportion of patients who successfully receive TACE/HAIC, .adverse events.

ELIGIBILITY:
Inclusion Criteria:

* HCC with diagnosis confirmed pathologically or clinically
* Patients who need to receive TACE and/or HAIC, or have plans to undergo another treatment (3-6 weeks after the previous treatment)
* Child Pugh class A or B
* ECOG PS 0-2
* PLT ≤ 75×10^9/L (10 days before interventional therapy)

Exclusion Criteria:

* Thrombocytopenia caused by hematological diseases, non chemotherapy related thrombocytopenia (excluding liver cirrhosis with hypersplenism)
* PLT <30×10^9/L
* History of hepatic encephalopathy, refractory ascites, or hepatorenal syndrome
* History of arterial or venous thrombosis within 6 months
* Uncontrolled severe infections
* Pregnant or breastfeeding female patients
* Immune deficiencies, such as autoimmune diseases, HIV infected individuals, etc
* Anticoagulation or antiplatelet therapy witch cannot be suspended during the treatment period: heparin, warfarin, rivaroxaban, dipyridamole, non-steroidal anti-inflammatory drugs, aspirin, verapamil, Ticlopidine, clopidogrel, glycoprotein IIb/IIIa antagonists, erythropoietin, etc;
* Administration of blood products within 7 days prior to the baseline visit (excluding albumin infusion)
* Allergy to avatrombopag or any of its formulations
* History (such as gastrointestinal bleeding within 3 months, high risk of thrombosis, such as portal vein main flow velocity<10cm/s) which may affect the safety of the patients or their ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with PLT >75×10^9/L or doubling from baseline | 1 year
  The proportion of patients with PLT >75×10^9/L or doubling from baseline

SECONDARY OUTCOMES:
Proportion of patients with PLT >75×10^9/L | 1 year
  The proportion of patients with PLT >75×10^9/L
Proportion of patients with PLT doubling from baseline | 1 year
  The proportion of patients with PLT doubling from baseline
Increace in PLT | 1 year
  the Increace in PLT after treatment
Proportion of patients who successfully receive TACE/HAIC | 1 year
  The proportion of patients who successfully receive TACE/HAIC
Adverse events (AEs) | 1 year
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No